CLINICAL TRIAL: NCT07146828
Title: Clinical Application Research of 5-Degree (0.05 D) Precision Optometry in Corneal Refractive Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-K173
Record Dates: First submitted 2025-08-15; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Refractive Surgery
Keywords: Corneal refractive surgery; SMILE; FS-LASIK; 0.05 D precision refraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional group (No Intervention): The traditional group had their infusion rates based on past experience.
- 0.05 D refraction Group (Experimental): The 0.05 D refraction group had their infusion rates precisely calibrated using 0.05 D refraction by the Binocular Wavefront Optometry Machine (BWFOM, Ai-Zhitong Medical Technology Co., Ltd., Zhejiang, China)
  Interventions: Device: Binocular Wavefront Optometry Machine (BWFOM, Ai-Zhitong Medical Technology Co., Ltd., Zhejiang, China)

INTERVENTIONS:
Device: Binocular Wavefront Optometry Machine (BWFOM, Ai-Zhitong Medical Technology Co., Ltd., Zhejiang, China) — The 0.05 D refraction group had their infusion rates precisely calibrated using 0.05 D refraction by the Binocular Wavefront Optometry Machine
  Arms: 0.05 D refraction Group

SUMMARY:
In recent years, the incidence of myopia has been high globally and is exhibiting a rapid upward trend, with projections estimating it will reach 49.8% by 2050. Corneal refractive surgery has become a primary method for correcting myopia, demonstrating significant efficacy and favorable safety. However, studies indicate that overcorrection or undercorrection can occur following refractive surgery. Reports have shown that three months post-SMILE surgery, 20% of eyes had residual refractive errors ≥ 0.50 D, and 6% had errors ≥ 1.00 D. We hypothesize that this may be related to imprecise preoperative refraction, subsequently affecting postoperative visual quality.

Due to limitations in lens manufacturing precision, the widely used increment for sphere correction remains 0.25 D. However, this may prevent some patients from achieving their optimal corrected state. Studies have reported that 95% of individuals are sensitive to diopter changes below 0.25 D, and 44% can distinguish changes smaller than 0.125 D. Other research suggests that adjusting spherical power in 0.05 D increments yields better corrected visual acuity. Furthermore, scholars have reported that 0.05 D precision refraction can significantly improve the red-green balance test rate, enabling myopic patients to achieve better visual quality. Therefore, improving refraction precision could provide patients with superior visual outcomes.

Currently, the Binocular Wavefront Optometry Machine (BWFOM, Ai-Zhitong Medical Technology Co., Ltd., Zhejiang, China) can perform objective and subjective refraction with 0.05 D increments for both sphere and cylinder correction, while also separately measuring higher-order aberrations (HOAs) and lower-order aberrations (LOAs). Given the scarcity of research on the outcomes of 0.05 D refraction for SMILE and FS-LASIK procedures, this study aims to evaluate visual acuity, aberrations, and refractive status in patients following SMILE and FS-LASIK surgery. The primary objective is to investigate whether preoperative 0.05 D precision refraction using the BWFOM can enhance postoperative visual quality for SMILE and FS-LASIK patients.

DETAILED DESCRIPTION:
This study aims to optimize the surgical parameters of corneal refractive surgery (SMILE and FS-LASIK) by utilizing 0.05 D high-precision refraction achieved through a binocular wavefront aberrometer, thereby improving patients' postoperative visual outcomes. The prospective study design involves patients scheduled for corneal refractive surgery at our hospital.

The research consists of two parts:

Part One: Performing 0.05 D precision refraction on myopic patients using the binocular wavefront aberrometer.

Part Two: Applying the obtained refraction results (in increments of 0.05 D) for refractive correction in patients undergoing SMILE and FS-LASIK surgery.

Specific procedures include:

Screening eligible patients who voluntarily choose SMILE or FS-LASIK. Preoperatively inputting the patients' 0.05 D refraction data into the SMILE platform (VisuMax Precision 4.0 - VISULYZE system) or the FS-LASIK system (applying the manufacturer-provided nomogram for undercorrection).

Utilizing the system-recommended input values for correcting refractive errors during surgery.

Conducting postoperative follow-up examinations at 10 days, 1 month, 3 months, 6 months, and 1 year.

Evaluation metrics include:

1. Primary Endpoint Indicators:

   Postoperative uncorrected visual acuity (UCVA), best-corrected visual acuity (BCVA), spherical power, cylindrical power, spherical equivalent (SE), and aberrations.

   Proportion of patients achieving postoperative UCVA ≥ 0.8, ≥ 1.0, and ≥ 1.2. Proportion of patients with postoperative SE within ±0.50 D and ±1.0 D. Proportion of patients with postoperative astigmatism (cylinder) within ±0.50 D and ±1.0 D.

   Postoperative efficacy index and safety index.
2. Safety Indicators:

Intraocular pressure (IOP). Anterior segment examination.

ELIGIBILITY:
Inclusion Criteria:

1. The diopter is relatively stable (the diopter increases within -0.50D per year for 2 consecutive years);
2. Age: 18 to 40 years old;
3. Optimal preoperative corrected visual acuity >= 4.8;
4. More than 2 weeks for soft contact lenses and more than 3 months for hard contact lenses before surgery
5. Patients who are willing to perform SMILE surgery

Exclusion Criteria:

1. Patients with history of eye surgery and trauma;
2. Patients with keratoconus tendency;
3. systemic connective tissue diseases and autoimmune diseases;
4. Patients with high blood pressure, diabetes and heart disease history;
5. Other eye disease history such as uveitis, scleritis and other eye inflammation patients;
6. Patients with scar constitution.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative spherical equivalent | Preoperatively, and at 1 day, 10 days, 1 month, 3 months, 6 months, and 1 year postoperatively
  It calculated as: SE = Sphere + ½ Cylinder
Postoperative corrected distance visualacuity | Preoperatively, and at 1 day, 10 days, 1 month, 3 months, 6 months, and 1 year postoperatively
  Using the standard logarithmic visual acuity chart, with units in logMAR.
Postoperative uncorrected distance visual acuity | Preoperatively, and at 1 day, 10 days, 1 month, 3 months, 6 months, and 1 year postoperatively
  Using the standard logarithmic visual acuity chart, with units in logMAR
spherical diopter | Preoperatively, and at 1 day, 10 days, 1 month, 3 months, 6 months, and 1 year postoperatively
  Spherical diopter (D) is the unit of measurement for the refractive (light-bending) power of a spherical lens (or the spherical component of a corrective lens) used to correct myopia (nearsightedness) or hyperopia (farsightedness).
cylinder diopter | Preoperatively, and at 1 day, 10 days, 1 month, 3 months, 6 months, and 1 year postoperatively
  The unit of measurement for the lens power required to correct astigmatism, representing the difference in refractive power between the steepest and flattest meridians (axes) of the eye or lens

CONTACTS AND LOCATIONS:
Locations (1):
- Binocular Wavefront Optometry Machine, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No